# An Observational Study: Investigating Participation Patterns of Patients in Atopic Dermatitis Clinical Trials

# An Informed Consent Form For Power Clinical Trial's Observational Clinical Study

Date: December 8, 2023

#### About This ICF - An Introduction

This brief summary aims to provide an overview of our observational clinical study, emphasizing its procedures, potential risks, and benefits for participants. Your consent is a requirement, but participation is entirely voluntary. You possess the right to withdraw at any time without facing any repercussions.

Our study endeavors to comprehend why patients with atopic dermatitis opt to join, continue, or withdraw from clinical trials. The primary procedures involve completing questionnaires and follow-up calls, structured to minimize any potential risks to participants.

While participants may not experience direct medical benefits in this observational study, the collected data will serve to identify methods for enhancing clinical trial participation rates, ultimately benefiting those with atopic dermatitis.

The study's findings will furnish valuable insights into the factors influencing clinical trial participation rates. Our aim is to refine recruitment strategies and increase patient engagement in trials, leading to better treatment options and outcomes for atopic dermatitis patients. Nonetheless, participation in this study is voluntary, and declining won't impact your rights or privileges.

Carefully reviewing the consent form and seeking clarification on any concerns before making a decision is crucial. Engaging with family, friends, advisors, and healthcare professionals for discussions is also recommended to ensure an informed choice.

Your participation is entirely voluntary, and you possess the right to withdraw at any time without any consequences.

Understanding Participation Factors in Atopic Dermatitis Clinical Trials

Clinical trials serve a crucial role in advancing atopic dermatitis treatments. Yet, questions arise about whether trial participants truly represent the wider population. This trial aims to delve into what influences patients regarding enrollment, discontinuation, or resumption in atopic dermatitis clinical trials. Grasping these factors will enhance future study relevance and effectiveness.

To ensure robust findings, we aim to recruit a diverse demographic range. Exploring factors like age, race, income, and education's impact on participation decisions is pivotal. Gathering this data aims to devise improved strategies for engaging underrepresented groups in future clinical trials.

Participation in this trial is voluntary, allowing individuals to withdraw anytime without repercussions. The study involves minimal risk through questionnaire completion and follow-up calls. Prospective participants are strongly urged to review the consent form thoroughly and ask any clarifying questions.

In essence, this trial aims to deepen our comprehension of factors affecting atopic dermatitis clinical trial participation. Augmenting participation rates can expedite the development of innovative treatments for this debilitating disease.

Examining Atopic Dermatitis Patient Participation in Clinical Trials

Our observational clinical research endeavors to understand the factors influencing atopic dermatitis patients in their choices regarding clinical trial participation—enrollment, withdrawal, and completion. Seeking participants from ongoing or past interventional trials, we'll identify potential participants using electronic medical records.

Upon opting in, our staff will provide a consent form, elucidating the study's objectives and participant rights. Data collection involves biweekly questionnaires on demographics, medical history, and reasons guiding trial participation. Additionally, quarterly phone or video interviews will be conducted for in-depth insights.

Statistical analysis of gathered data aims to uncover the variables shaping patient participation. Sharing findings through conferences and scholarly publications aims to benefit stakeholders in clinical trials.

Our discoveries aim to enhance future clinical studies for atopic dermatitis patients by bolstering recruitment and retention.

Participation is entirely voluntary, allowing withdrawal at any time sans consequences. Minimal risks include questionnaire completion and follow-up interviews. Queries or concerns can be addressed by our accessible research team.

Assessing Risks in Atopic Dermatitis Observational Studies

Observational clinical research studies focusing on atopic dermatitis do not involve experimental treatments, yet participation may carry potential risks. These risks might involve privacy breaches, emotional distress due to the study's subject matter, and potential negative outcomes from trial-related procedures.

Prior to participation, it's crucial to meticulously review and comprehend the informed consent form and address any concerns with the research team. The team will offer detailed insights into potential risks, study benefits, and safety measures implemented to safeguard participants' well-being.

Understanding the Potential Benefits of Atopic Dermatitis Observational Trials

Participating in observational clinical trials for atopic dermatitis offers patients a chance to contribute to medical advancements and potentially enhance future treatment options. Despite lacking experimental therapies, patients can still receive attentive care during the study period.

Prior to deciding on trial participation, patients should meticulously assess potential benefits and risks based on their individual situation and goals. Consulting healthcare providers and the research team is crucial in making an informed decision.

Considerations Leading to the Conclusion of Your Participation

Realizing that your participation in a clinical trial can be halted without your consent holds significance. Researchers or sponsors may terminate it due to reasons like study suspension, funding withdrawal, or if it's deemed beneficial for you.

Furthermore, your involvement might cease due to declining health, pregnancy, opting out post-notification of impactful changes, or non-compliance with study guidelines. Carefully reflecting on these elements before committing to a clinical trial is crucial.

Atopic Dermatitis Clinical Trials: A Comparative View

In atopic dermatitis clinical trials, participation is completely optional, granting the right to withdraw without adverse consequences.

For a global view of <u>atopic dermatitis studies</u>, clinicaltrials.gov, managed by the National Institutes of Health (NIH), serves as a comprehensive trials database. Tailoring your search by location and medical condition is possible.

Furthermore, Power's reference page presents an updated list of currently recruiting atopic dermatitis trials.

Online Avenues to Explore Clinical Trial Diversity

Numerous online resources cater to individuals interested in understanding clinical trial diversity. Here are a couple of articles that might catch your attention:

Reid, Michel M., Scott P. Davis, Ouzama N. Henry, Ashwin A. Mathew, Scott McCallister, Taj T. Nero, Sanjit A. Rabheru, Shani H. Sampson, Tracy F. Vanderslice, and Danae T. Williams. "Demographic diversity of US-based participants in GSK-sponsored interventional clinical trials." *Clinical Trials* 20, no. 2 (2023): 133-144.

Lund, Mary Jo, Mark T. Eliason, Ann E. Haight, Kevin C. Ward, John L. Young, and Rebecca D. Pentz. "Racial/ethnic diversity in children's oncology clinical trials: ten years later." *Cancer: Interdisciplinary International Journal of the American Cancer Society* 115, no. 16 (2009): 3808-3816.

These websites offer valuable information on the challenges surrounding clinical trial diversity and the proposed solutions.

## **Ensuring Privacy in Research Studies**

The confidentiality of the personal information collected for this research is a top priority. While complete confidentiality cannot be guaranteed at all times, extensive measures have been taken to protect it. Note that legal obligations might necessitate the disclosure of personal information. However, no research publications or presentations will disclose your name or personally identifying information.

Various entities, including accrediting bodies, government regulatory authorities (such as the FDA and OHRP), safety monitors, study sponsors, and authorized representatives, may access your medical information for research, quality assurance, and data analysis purposes.

In rare cases, we might request an "Authorization Form" outlining the use and sharing of your information for this study. Before sharing your information or research samples with Power researchers, other university institutions, or external commercial firms for future research, explicit consent will be obtained. Your confidential data will be securely handled and removed.

### Agreement to Informed Consent Terms

Your signature on this consent agreement signifies your acknowledgment and acceptance of the following:

- You have comprehensively read and understood this informed consent form, with encouragement to seek alternative viewpoints before decision-making.
- All your queries concerning the research project and its methodologies have been satisfactorily answered, equipping you with the necessary information for study participation.

- Consideration has been given to potential benefits, drawbacks, and alternatives related to participation in the research.
- Your voluntary involvement in the research study will not restrict your ability to exercise your legal rights.
- Any significant updates impacting your decision to continue participating in the research study will be promptly communicated to you.
- This consent form has been provided, offering you the opportunity to address any questions you might have had.

| Participant's Signature | | |
|---|---|---|
| Name of Participant | Signature of Participant | Date |
| Confirmation by the Researcl | her | |
| As the researcher, I have taken th adequately and provide a comprehave verified that the patient's par consent. | hensive understanding of the stu | dy. Furthermore, I |
| Signature of Researcher Who | o Received Consent | |
| Name of Investigator | Signature of Investigator | <br>Date |